CLINICAL TRIAL: NCT00848159
Title: Evaluation of Thoracic Kyphosis in Elderly Women Affected by Osteoporosis Through Computerized Photogrammetry
Brief Title: Postural Assessment by Photogrammetry
Status: Completed | Type: Observational
Sponsor: Universidade de Franca (Other)
Responsible Party: Lislei Jorge Patrizzi, Universidade de Franca
Other Study IDs: 041/07
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; kyphosis; photogrammetry
MeSH Terms: conditions — Osteoporosis; Kyphosis

STUDY DESIGN:
Biospecimen Retention: The two groups were photographed in the sagittal plane with right column markers fixed on two anatomical points. The selected images were quantified by computerized photogrametry, using the program Autocad-2006
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Group 1 was composed of six women with a densitometric diagnosis of osteoporosis in column (DP =- 2.70 to -4.97), with an average weight of 57.5 (+6.9) kg, mean height of 1 , 4 (+ 0.07) my body mass index (BMI) of 26.1 (+1.8) Kg/m2
- 2: Group 2 consists of six women with a densitometric diagnosis of osteopenia in column (DP =- 1.07 to -2.09), with an average weight of 62.1 (+9.9) kg, mean height of 1, 5 (+0.03) I BMI 25.3 (3.3) kg/m2, both compared with young adults

SUMMARY:
This study aimed to measure the degree of thoracic kyphosis in elderly women with those affected by osteoporosis in the spine, through photogrammetry computer and check the difference between the values obtained with the assumption of greater thoracic kyphosis in osteoporotic women.

DETAILED DESCRIPTION:
The decrease in bone density of vertebrae leads to a reduction of the anterior vertebral bodies, resulting in compression and collapse of vertebrae, with narrowing of intervertebral disc spaces and, determining a number of deformities in the spine and postural changes, among which can highlight the increase in thoracic kyphosis. This becomes significantly higher with age and after menopause, defined as an increase in curvature in the sagittal plane of the thoracic spine.

Radiographic images have been used for the measurement of thoracic kyphosis, but with some drawbacks of this method such as radiation exposure, radiographic image quality unsatisfactory hampering its analysis and the lack of equipment in the physical environment to monitor clinical evolution of the treatment, causing thus the search for noninvasive methods for evaluating the curves of the spine, including the photogrammetry computed.

According to the American Society of Photogrammetry, the computed photogrammetry is "the art, science and technology of information on physical objects and environment through processes of recording, measuring and interpreting photographic images and patterns of electromagnetic radiant energy and other sources." It is a widely used tool for assessment by quantifying the postural changes through the application of photogrammetric principles to photographic images obtained in body movements, adding to the diagnostic evaluation for physical therapy in different areas.

ELIGIBILITY:
Inclusion Criteria:

* age between 50 and 80 years
* with examination of bone densitometry
* with densitometric diagnosis of osteopenia in the first group, the second group for osteoporosis,
* willing to participate in the study

Exclusion Criteria:

* presence of severe scoliosis, ankylosing spondylitis, obesity
* presence of neurological diseases serious

Ages: 65 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The investigators evaluated 12 women with mean age of 68.5 years (range 65 to 74 years), divided into two groups. Group 1 consists of six women with a densitometric diagnosis of osteoporosis in column (SD: -2.70 to -4.97) and group 2 consists of six women with a densitometric diagnosis of osteopenia in column (DP: 1.07 to -2 , 09), both compared with young adults.
Sampling Method: Non-Probability Sample
Enrollment: 12
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Computerized Photogrammetry

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cristina Rodrigues, Principal Investigator — Universidade de Franca; Lislei Patrizzi, Principal Investigator — Universidade de Franca